CLINICAL TRIAL: NCT05217095
Title: Clinical Trial on a Novel Blood Pumping System in 4008A Hemodialysis Machine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: D.med Consulting GmbH (Industry)
Collaborators: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: D.Med 20-01 Convergence
Record Dates: First submitted 2021-12-13; First posted 2022-02-01 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Renal Dialysis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional Group (Other): Each patient will be treated for one session of dialysis after enrolled. Each of them will have only one treatment in the middle of the week (Wednesday or Thursday). The patients will be treated using 4008A dialysis machines in combination with a sidecar and the convergence dialyzer as investigational devices.Each patient will be treated according their regular treatment and laboratory analysis will be taken. The blood level of free hemoglobin ( fHb ) will be taken on 30 min by use of HemoCue device. ACT time will be measured on 15 min and for that 0.5 ml blood from venous line will be taken.
  Interventions: Device: Convergence Dialyzer

INTERVENTIONS:
Device: Convergence Dialyzer — The Convergence dialyzer with design changes made to FX Coral 600 dialyzer will be tested together with Sidecar. In the dialyzer is integrated centrifugal-flow blood pump.The centrifugal-flow blood pump replaces the peristaltic roller pump of the extracorporeal circuit which pumps blood from patient to the dialyzer and from dialyzer to the patient. The centrifugal-flow blood pump is designed to transport blood from the patient to the dialyzer, and after purification, return the blood to patient.

SUMMARY:
The aim of this clinical trial will be to verify the feasibility of using an impeller system instead of a roller pump for hemodialysis, using the established 4008 hemodialysis system and a Convergence Dialyzer with design changes made to the FX-Coral P 600 dialyzer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be up to 18-85 years
* Hemodialysis Schedule: 3 times per week; app. 3- 5 hour treatment
* Stable clinical conditions: no recent (last 2 weeks) hospitalization events, no recent main surgery (last 3 weeks), no acute cardiological problems, hemoglobine levels in the DOQI Guideline ranges.
* Hemodynamic stability during dialysis i.c. number of sessions complicated by acute hypotension events or arrhythmia <25% in the last 3 Months
* Well-functioning AVF vascular access: access recirculation ≤10%
* No coagulation disorders and anticoagulant therapy
* Patients must be using a similar size dialyzer as Convergence dialyzer
* Signed Inform consent form.

Exclusion Criteria:

* Unstable clinical condition: recent hospitalization, recent surgery, anemia, active neoplastic diseases,shock or unstable cardiac function and intolerable to extracorporeal treatment
* Hemodynamic instability during the dialysis sessions; more than 25% of the sessions complicated by acute hypotension or arrhythmic events.Presence of clinically significant abnormality on a 12-lead ECG at Screening that, at the investigator's clinical judgment, may compromise the safety of the patient or affect the outcome of the study.
* History or presence of congestive heart failure with symptoms consistent with New York Heart Association Class III or IV functional status within 6 months prior to the study Convergence system treatment.
* Abnormal liver function values including but not limited to the aspartate transaminase, alanine transaminase or alkaline phosphatase ≥5 × upper limit normal.
* Any uncontrolled clinically significant respiratory disease in the investigator's opinion (e.g., chronic obstructive pulmonary disease, cystic fibrosis, bronchiectasis, asthma).
* Temporary excluded will be patients with increased body temperature due to some infective disease, dehydration, diarrhea, hyperglycemia,
* Severe bleeding, or history or evidence of bleeding diathesis or coagulopathy with the risk of bleeding or have to put on dialysis without anticoagulant.
* Using temporary or permanent dialysis catheter
* Uncontrolled diabetes mellitus or hypertension, at the discretion of investigator.
* Known pregnancy and lactating without pregnancy test
* Patient has known allergy or hypersensitivity reaction to dialyzer membrane or other disposable
* Any conditions significantly affecting the nervous system (i.e., neuropathic conditions or nervous system damage
* Patient shows evidence of a condition (psychological, emotional problems, any disorders or resultant therapy) that is likely to invalidate health information, consent, or limit the ability of the patient to comply with the protocol requirements in the opinion of the investigator
* Any other conditions at the discretion of investigator not suitable for patients to participate in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-01-22 (Actual); Study Completion 2022-02-22 (Actual)

PRIMARY OUTCOMES:
Incidence of Alarms | 1 study day
  Incidence of alarms leading to end of treatment, cause identification
Product defects | 1 study day
  Product defects leading to end of treatment, cause identification
Serious adverse event / adverse event/ Serious adverse device effect/ Adverse device effect/Unanticipated serious adverse device effect | 1 study day
  Incidence of Serious adverse event / adverse event/ Serious adverse device effect/ Adverse device effect/Unanticipated serious adverse device effect
Incidence of "recoverable" alarms | 1 study day
  Incidence of "recoverable" alarms, cause of alarms i.e.arterial/venous pressure outside of set range/limits

SECONDARY OUTCOMES:
Completion Rate | 1 study day
  The completion rate of a dialysis session according to prescription. The study is considered to be successful, if at least 8 patients reach the effective dialysis time.
Average Blood Flow Rate | 1 study day
  The average blood flow rate is measured during the dialysis treatment. Maintenance of preset blood flow rates throughout the dialysis in at least 8 out of 10 patients
Arterial pressure | 1 study day
  The arterial pressure is measured in mmHg.
Venous pressure | 1 study day
  The venous pressure is measured in mmHg.
Impeller RPM | 1 study day
  The rotation of the impeller pump is measured in rpm.
Dialysis Dose as single pool Kt/V | 1 study day
  The delivered dialysis dose as single-pool Kt/V. Achievement of a spKt/V > 1.4 in at least 8 out of 10 patients.
Dialysis Dose as Urea Reduction Ratio (URR) | 1 study day
  The delivered dialysis dose as URR.
Ultrafiltration Volume | 1 study day
  Total ultrafiltration volume (ml). Achievement of preset total ultrafiltration volume (ml) to reach dry weight target in at least 8 out of 10 patients.
Body weight change | 1 study day
  Patient body weight change (before treatment vs. after treatment).
pH | 1 study day
  The blood level of pH is measured pre/post HD. Achievement of results in laboratory acceptable ranges,
Bicarbonate | 1 study day
  The blood level of Bicarbonate is measured pre/post HD. Achievement of results in laboratory acceptable ranges.
Potassium | 1 study day
  The blood level of Potassium is measured pre/post HD. Achievement of results in laboratory acceptable ranges,
Sodium | 1 study day
  The blood level of Sodium is measured pre/post HD. Achievement of results in laboratory acceptable ranges.
Chloride | 1 study day
  The blood level of Chloride is measured pre/post HD. Achievement of results in laboratory acceptable ranges.
Free hemoglobin | 1 study day
  The blood level of free hemoglobin (fHb measured on 30 min) to be in acceptable ranges for hemolysis
Anticoagulation | 1 study day
  The total dose of anticoagulation consumption not to exceed patient treatment dose as I.U per kg
Clotting Score | 1 study day
  The clotting score of dialyzer(visual check, using common scale for dialyzer study)
  1. No visible thrombosed fibers
  2. A few visible thrombosed fibers
  3. Moderately visible thrombosed fibers
  4. Many visible thrombosed fibers
  5. Completely visible thrombosed fibers
  So the score goes from 1 (good) to 5 (bad).

CONTACTS AND LOCATIONS:
Overall Officials: Elena Babalj-Banskolieva, Dr., Principal Investigator — Specialized Hospital for Nephrology and Dialysis Diamed
Locations (1):
- Special Hospital for Nephrology and Dialysis Diamed, Skopje, North Macedonia

IPD SHARING:
Plan to Share IPD: No